CLINICAL TRIAL: NCT05594082
Title: Real-world Effectiveness and Safety Study of T-Dxd in Chinese Metastatic Breast Cancer.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-24
Record Dates: First submitted 2022-10-08; First posted 2022-10-26 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Trastuzumab Deruxtecan, 5.4 mg/kg ivgtt q3w

SUMMARY:
The aim of this trial is to explore the real-world effectiveness and poteintial predictors in Chinese metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old.
2. Metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
3. Plan to receive or has received Trastuzumab Deruxtecan monotherapy
4. Available medical history.

Exclusion Criteria:

1. Incomplete medical history.
2. Pregnancy or breast-breeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese metastatic breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  progression-free survival

SECONDARY OUTCOMES:
ORR | 6 weeks
  Overall Response Rate
CBR | 6 weeks
  Clinical benefit Rates
OS | 6 weeks
  Overall Survival
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China